CLINICAL TRIAL: NCT00566709
Title: Phase II Study of Usefulness of Near Infrared Spectroscopy to Optimize Red Blood Cells Transfusion in Neuro Critical Ill Patients With Severe Traumatic Brain Injury, Subarachnoid Hemorrhage or Intracerebral Hemorrhage.
Brief Title: Near Infrared Spectroscopy (NIRS) as Transfusion Indicator in Neurocritical Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Santiago R. Leal-Noval, Santiago R. Leal-Noval, MD Ph.D, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-0157/2006; PI 157/06
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage; Intracerebral Hemorrhage
Keywords: transfusion; NIRS; cerebral oxygenation; red blood cell; near infrared spectroscopy
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RBCT based on rSO2 value (Experimental): Intervention: In the rSO2 - strategy group, patients will be transfused to attain a post-transfusion rSO2 values higher than 60%.
  Interventions: Procedure: Red blood cells transfusion
- RBCT based on hemoglobin level value (Active Comparator): Intervention: In the hemoglobin - strategy group, patients will be transfused to reach post-transfusion hemoglobin levels between 8.5 g/dL and 10 g/dL.
  Interventions: Procedure: Red blood cells transfusion

INTERVENTIONS:
Procedure: Red blood cells transfusion — Patients will be transfused (one to one red blood cells unit transfusion)

SUMMARY:
Neurocritical ill patients are frequently transfused. Red blood cell transfusion (RBCT) in these patients has been associated with deleterious effects, including higher rates of nosocomial infections, multi-organ failure, and mortality. Therefore, it seems crucial to avoid any unnecessary RBCT.

Most critically ill patients tolerate hemoglobin levels near 7 g/dL without an increase in morbidity or mortality rates. In this regard, a recent sub-analysis of TRICC trial has showed that TBI patients may tolerate hemoglobin levels as low as 7 g/dL, but other studies including neurocritical patients suggested that severe anemia may worsen clinical outcome. Therefore, optimal hemoglobin levels in neurocritical care patients remain largely unknown. Some textbooks and guidelines recommend to transfuse these patients to reach hemoglobin levels near to 10 g/dL, despite the lack of a solid scientific background supporting this target.

Even though it has not been demonstrated, hemoglobin-based RBCT prescription could result in over- or under-transfusion in neurocritical patients. Alternatively, it has been suggested that more physiological transfusion triggers, using direct signals coming from the brain, will progressively replace arbitrary hemoglobin-based transfusion triggers in the neurocritical patients [65]. At the neurocritical units, patients are often monitored by using non-invasive methods, such as near infrared spectroscopy which indirectly measures regional cerebral oxygen saturation (rSO2). Changes in rSO2 values have been shown to directly correlate with changes in erythrocyte mass, thus increasing with RBCT and decreasing with blood losses. Moreover, rSO2 values also show a good correlation with clinical outcome and other variables which are often monitored in TBI patients.

The purpose of this study is to ascertain as to whether rSO2 levels are more efficacious than conventional hemoglobin levels in guiding RBCT in patients admitted to a neurocritical care unit.

ELIGIBILITY:
Inclusion Criteria:

* Severe traumatic brain injury (Glasgow coma scale < 9), subarachnoid hemorrhage (Hunt and Hess scale ≥ 3) or intracranial hemorrhage
* Moderate anemia. Hemoglobin levels > 7 g/dL and < 10 g/dL
* Hemodynamical stability (mean arterial pressure > 75 mm Hg)
* Respiratory stability (PaO2 / FiO2 ratio > 220)
* Expected length of ICU stay > 3 days

Exclusion Criteria:

* Patient's relatives' refusal to patient's inclusion in the study
* Active bleeding
* Ongoing need for blood products
* Patients necessitating ongoing resuscitation
* End-stage in which death is imminent
* Antecedents of angina or myocardial infarction (poor cardiopulmonary reserve)
* Deficient signal of rSO2 impeding its proper valuation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago R Leal-Noval, MD, PhD, Principal Investigator — Hospital Universitario "Virgen del Rocío", Seville, Spain; Victoria Arellano, MD, PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Rosario Amaya, MD, PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Antonio M Puppo, MD, PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Carmen M Ferrándiz, MD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Antonio J Marín, MD, PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Francisco Murillo, MD, PhD, Study Director — Hospital Universitario "Virgen del Rocío", Seville, Spain; Manuel Muñoz, Prof, MD, PhD, Study Chair — Prof Transfusion Medicine University of Malaga, Spain; Vicente Padilla, MD, Study Chair — Hospitales Universitarios Virgen del Rocío; Yael Corcia, MD, Study Chair — Hospitales Universitarios Virgen del Rocío; Aurelio Cayuela, MD, PhD, Study Chair — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario "Virgen del Rocío", Seville, Seville, Spain

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Leal-Noval SR, Arellano-Orden V, Munoz-Gomez M, Cayuela A, Marin-Caballos A, Rincon-Ferrari MD, Garcia-Alfaro C, Amaya-Villar R, Casado-Mendez M, Dusseck R, Murillo-Cabezas F. Red Blood Cell Transfusion Guided by Near Infrared Spectroscopy in Neurocritically Ill Patients with Moderate or Severe Anemia: A Randomized, Controlled Trial. J Neurotrauma. 2017 Sep;34(17):2553-2559. doi: 10.1089/neu.2016.4794. Epub 2017 Jul 19. PMID 28486023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Started | 51 | 51
Completed | 46 | 51
Not Completed | 5 | 0
Not completed — Protocol Violation | 5 | 0

BASELINE CHARACTERISTICS:
Population: Patient included into to "Intention to treat" analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (18.3) | 46.1 (16.3) | 45.6 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 35 | 31 | 66
Hemoglobin (g/L) [Mean (Standard Deviation); unit: g/L] | 110.9 (21.2) | 114 (21.6) | 112.4 (21.3)
Arterial Hypertension (n) [Number; unit: participants]
  Yes | 14 | 15 | 29
  No | 37 | 36 | 73
Diabetes mellitus (n) [Number; unit: participants]
  Yes | 2 | 5 | 7
  No | 49 | 46 | 95
APACHE II score [Mean (Standard Deviation); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation (APACHE) II score Minimun score:0, Maximum score: 71 Higher values represent worse result.
  units on a scale | 14.6 (4.8) | 13.8 (4.2) | 14.1 (4.5)
GCS [Median (Inter-Quartile Range); unit: units on a scale] — Glasgow Coma Scale Minimun: 3; Maximum: 15 Higher values represent better outcome
  units on a scale | 9 [7 to 12] | 9 [7 to 11] | 9 [7 to 11]
ISS score (N=30, 27) [Mean (Standard Deviation); unit: units on a scale] — Injury severity score (ISS) Minimum: 0; maximum: 75 Higher values represent worse outcome
  ISS is only collected in patients with traumatic brain injury (N=57)
  * 30 into rSO2 arm
  * 27 into hemoglobin arm
  units on a scale | 28.0 (9.8) | 29.0 (9.6) | 28.5 (9.6)
Hunt and Hess scale (N=10, 13) [Mean (Standard Deviation); unit: units on a scale] — Hunt and Hess scale for assessing the severity of patients with subarachnoid hemorrhage Minimum: 1; Maximum: 5 Higher values represent worse outcome
  Only 23 patients with subarachnoid hemorrhage are included.
  * 10 into rSO2 arm
  * 13 into hemoglobin arm
  units on a scale | 4.1 (1.2) | 4.1 (0.8) | 4.1 (1)
Fisher scale (N=10, 13) [Mean (Standard Deviation); unit: units on a scale] — Computer tomography Fisher Scale
  Minimum: 1; Maximum: 4
  Higher values represent worse outcome
  Only 23 patients with subarachnoid hemorrhage are included
  * 10 into rSO2 arm
  * 13 into hemoglobin arm
  units on a scale | 3.9 (0.3) | 3.8 (0.4) | 3.8 (0.4)
Modified Grab score (N=11, 11) [Mean (Standard Deviation); unit: units on a scale] — Modified Graeb score for intra cerebral hemorrhage Minimum: 0; maximum: 42.
  Higher values represent worse outcome
  Only 22 patients with intra cerebral hemorrhage are included
  * 11 into rSO2 arm.
  * 11 into hemoglobin arm.
  units on a scale | 6.7 (3.9) | 5.9 (3) | 6.3 (3.4)
PbrO2 (mm Hg) (N=17, 22) [Mean (Standard Deviation); unit: mm Hg] — Pressure brain regional oxygen: PbrO2
  Only 39 patients monitored with a PbrO2 probe are included:
  * 17 into rSO2 arm
  * 22 into hemoglobin arm
  mm Hg | 21.9 (5.7) | 22.8 (5.6) | 22.4 (5.6)
CPP (mm Hg) (N=17, 22) [Mean (Standard Deviation); unit: mm Hg] — Cerebral perfusion pressure (CPP)
  Only 39 patients monitored with a PbrO2 probe are included:
  * 17 into rSO2 arm
  * 22 into hemoglobin arm
  mm Hg | 73.9 (18.5) | 72.9 (15.6) | 73.4 (16.7)
Diagnosis [Number; unit: participants]
  Traumatic Brain Injury | 30 | 27 | 57
  Subarachnoid hemorrhage | 10 | 13 | 23
  Intra cerebral hemorrhage | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Units of Packed Red Blood Cell Transfused
Description: Number of units of packed packed red blood cell transfused, over the period that the patient was included into the protocol
Time Frame: duration of the protocol, an average of 15 days
Measure: Mean (Standard Deviation); unit: units
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Number analyzed (Participants) | 46 | 51
units | 0.9 (1.1) | 1.5 (1.4)
Statistical Analysis 1: Comparison: RBCT Based on rSO2 Value vs RBCT Based on Hemoglobin Level Value; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

2. Primary Outcome: Percentage of Transfused Patients in Each Group
Time Frame: duration of the protocol, an average of 15 days
Measure: Number; unit: percentage of transfused participant
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Number analyzed (Participants) | 46 | 51
percentage of transfused participant | 54.3 | 70.5
Statistical Analysis 1: Comparison: RBCT Based on rSO2 Value vs RBCT Based on Hemoglobin Level Value; Test type: Superiority or Other; p = 0.07, Chi-squared, Corrected

3. Secondary Outcome: Hospital Mortality
Time Frame: length of the hospital stay, an average of 20 days
Measure: Number; unit: participants
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Number analyzed (Participants) | 46 | 51
participants | 3 | 5
Statistical Analysis 1: Comparison: RBCT Based on rSO2 Value vs RBCT Based on Hemoglobin Level Value; Test type: Superiority or Other; p = 0.56, Chi-squared, Corrected

4. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Time Frame: The length of ICU stay, an avarege of 17 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Number analyzed (Participants) | 46 | 51
days | 21.00 (10.23) | 20.41 (11.06)
Statistical Analysis 1: Comparison: RBCT Based on rSO2 Value vs RBCT Based on Hemoglobin Level Value; Test type: Superiority or Other; p = 0.79, t-test, 2 sided

5. Secondary Outcome: Long-term Mortality
Time Frame: 1-year after hospital discharge
Measure: Number; unit: participants
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Number analyzed (Participants) | 46 | 51
participants | 12 | 12
Statistical Analysis 1: Comparison: RBCT Based on rSO2 Value vs RBCT Based on Hemoglobin Level Value; Test type: Superiority or Other; p = 0.77, Chi-squared, Corrected

6. Secondary Outcome: Unfavorable Glasgow Outcome Scale (GOS)
Description: GOS measures the degree of disability associated with the brain injury
  Unfavorable GOS included the categories of:
  1. death.
  2. vegetative status.
  3. severe disability.
Time Frame: At hospital discharge, an average of 21 days
Measure: Number; unit: participants
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Number analyzed (Participants) | 46 | 51
participants | 27 | 36
Statistical Analysis 1: Comparison: RBCT Based on rSO2 Value vs RBCT Based on Hemoglobin Level Value; Test type: Superiority or Other; p = 0.22, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: From admission of the patients into the protocol to the hospital discharge, an avarage 21 days
Arm/Group | RBCT Based on rSO2 Value | RBCT Based on Hemoglobin Level Value
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

LIMITATIONS AND CAVEATS:
Limited adherence to the protocol in the rSO2 arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No